CLINICAL TRIAL: NCT03888092
Title: A Phase Ib, Multi-center, Open-label Study of Z650 in Advanced Esophageal Squamous Cell Carcinoma (ECSS) With Epidermal Growth Factor Receptor (EGFR) Over Expression or Gene Amplification
Brief Title: Z650 in Advanced Esophageal Squamous Cell Carcinoma With EGFR Over Expression or Gene Amplification
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCD-DZ650-17-001
Record Dates: First submitted 2019-03-18; First posted 2019-03-25 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2022-05

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Z650 , Single-arm (Experimental): Z650 will be administered daily, at dose of 350 mg orally
  Interventions: Drug: Z650

INTERVENTIONS:
Drug: Z650 — receive oral Z650 once daily until disease progression or unacceptable toxicity occurs, each cycle is defined as 28 days
  Other Names: Larotinib

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Z650 in Advanced Esophageal Squamous Cell Carcinoma patients With EGFR Over expression or Gene Amplification.

DETAILED DESCRIPTION:
It is a multi-center , open-label, singer arm study to explore the safety and efficacy of Z650 in advanced ESCC patients who had experienced systematic chemotherapy. Approximately 45 subjects will be enrolled, each subjects will receive oral Z650, at dose of 350 mg/d, repeatedly until disease progression or unacceptable toxicity occurs, each cycle is defined as 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed Stage IIIB or IV ESCC
* At least experienced one regimens of chemotherapy prior to study
* Histological or cytological evidence of EGFR overexpression or gene copy number increased
* Measurable disease according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)
* Toxicity recovered to NCI CTCAE v.4.03 Grade ≤1 from previous treatments (except alopecia)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Life expectancy of ≥ 12 weeks
* Adequate organ function
* Subject Consent
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all the pertinent aspects of the trial prior to performing this study.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Prior treatments
* EGFR targeted therapy, or major surgery within 4 weeks prior to study treatment
* Nitrosourea and mitomycin chemotherapy within 6 weeks prior to study treatment
* Had received any investigational agent from other clinical study within 4 weeks prior to study treatment or are currently participating in other clinical trials
* Gastrointestinal diseases that could affect the absorption of Z650, (e.g., serious swallowing obstruction, chronic diarrhea, bowel obstruction);
* Symptomatic, untreated or unstable central nervous system metastases (patient are only permitted if treated, asymptomatic and stable for at least 4 weeks prior to start of study treatment)
* History of interstitial lung disease
* Uncontrolled hypertension that require more than two anti-hypertensive agents to control, or systolic blood pressure (BP) >140mmHg or diastolic BP >90 mmHg before the first administration
* Doppler ultrasound evaluation of Left ventricular ejection fraction < 50%
* Male with QTc interval > 450 ms or female with QTc interval > 470 ms
* History of immunodeficiency, or other acquired or congenital immunodeficiency, or history of organ transplantation
* Any disease of the following bellowed within 6 months prior to administration:

Myocardial infarction, or unstable angina, coronary or peripheral artery bypass graft, congestive heart failure, or cerebrovascular events (including transient ischemic attack)

* Active infection of hepatitis B virus (HBV)/hepatitis C virus (HCV), or infection of Human immunodeficiency virus (HIV)
* Other malignancies within 5 years prior to enrollment, with the exception of carcinoma in situ of the cervix, basal or squamous cell skin cancer
* History of serious allergic reactions attributed to excipients of Z650, including mannitol, sodium carboxymethyl starch, aerosol, magnesium stearate and silicified microcrystalline cellulose
* Pregnant women, or patients not agree to use of effective contraceptions during the study or within 6 month after the study
* Any other reason the investigator considers the patient is not suitable to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events (AEs) as a measure of safety and tolerability | up to 4 weeks after last dose
  AEs assessment via monitoring changes in vital signs (e.g.body temperature, pulse rate, blood pressure, respiratory rate,etc.) and physical examinations(e.g.height, weight, BMI,etc.)
Number of patients with adverse events (AEs) as a measure of safety and tolerability | up to 4 weeks after last dose
  AEs assessment via monitoring changes in clinical laboratory parameters (e.g. levels of liver, kidney, and bone marrow function) and ECG (e.g. QTc Interval).

SECONDARY OUTCOMES:
Overall response rate (ORR) | up to approximately 24 months
  Overall response rate (ORR), defined as a partial response (PR) or complete response (CR) occurring at any point post-treatment according to Response Evaluation Criteria in Solid Tumors as assessed by RECIST v1.1
Disease Control Rate (DCR) | up to approximately 24 months
  DCR, proportion of patients with best overall response of CR, PR or stable disease (SD)
Duration of Response (DOR) | up to approximately 24 months
  DOR, defined as time from the first documented CR or PR to first documented progression or death due to any cause
Progression-free Survival (PFS) | up to approximately 24 months
  PFS, defined as time from date of treatment to disease progression or death due to any cause
Overall Survival (OS) | up to approximately 24 months
  OS, defined as time from date of treatment to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Xu, PHD, Principal Investigator — Chinese PLA General Hospital, the Fifth Medical Center
Locations (1):
- Chinese PLA General Hospital, the Fifth Medical Center, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu R, Liu L, Zhao C, Bai Y, Zheng Y, Zhang S, Li N, Yang J, Fan Q, Wang X, Zeng S, Zhang Y, Zhang W, Zhuang Y, Kang N, Jiang Y, Sun H, Xu J. Larotinib in patients with advanced and previously treated esophageal squamous cell carcinoma with epidermal growth factor receptor overexpression or amplification: an open-label, multicenter phase 1b study. BMC Gastroenterol. 2021 Oct 23;21(1):398. doi: 10.1186/s12876-021-01982-4. PMID 34688250